CLINICAL TRIAL: NCT06716099
Title: Clinical Characteristics and Outcome of Patients With Community Acquired Pneumonia
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rania Abdo saeed, Rania Abdo Saeed, Sohag University
Other Study IDs: Soh-Med-24-09-01MS
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Community Acquired Pneumonia (CAP)
Keywords: CAP; Pneumonia; clinical characteristics
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum , urine , blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the goal of this observational study is to evaluate the clinical characteristic and outcomes of patients with community-acquired pneumonia admitted to Sohag University Hospital.

the researcher will take medical history and clinical examination and investigations of participants .

the participants will visit the clinic after one month to be reevaluated again .

DETAILED DESCRIPTION:
Community acquired pneumonia is acute infection of the pulmonary parenchyma that occurs in the community in a patient who has not been hospitalized within 14 days prior to onset of symptoms or hospitalized less than 2 days prior to the onset of symptoms the aim of the study typically focuses on examining the various factors that influence the presentation, management, and outcomes of individuals diagnosed with pneumonia that is acquired outside of a hospital or healthcare setting.

Type of the study: observational study

Outcomes of interest include:

I. Mortality (in hospital and 30 days). II. The need for further mechanical ventilation or ICU admission. III. Duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients ≥18 years old with community acquired pneumonia

Exclusion Criteria:

1. Patients already was diagnosed as active malignancy before admission
2. Patient on chemotherapy
3. HIV patients
4. Indication of mechanical ventilation on admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: participants will be more than 18 years old who admitted to sohag university hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
improved | within one month
  when the patient is improved and discharged
patients developed complications | within one month
  when patients developed complications like acute kidney injury , septic shock or Disseminated intravascular coagulopathy
Death of patient | within one month

SECONDARY OUTCOMES:
intensive care unit admission | within one month

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Result] Han X, Liu X, Chen L, Wang Y, Li H, Zhou F, Xing X, Zhang C, Suo L, Wang J, Yu G, Wang G, Yao X, Yu H, Wang L, Liu M, Xue C, Liu B, Zhu X, Li Y, Xiao Y, Cui X, Li L, Cao B; CAP-China network. Disease burden and prognostic factors for clinical failure in elderly community acquired pneumonia patients. BMC Infect Dis. 2020 Sep 12;20(1):668. doi: 10.1186/s12879-020-05362-3. PMID 32919458
- [Result] Iqbal N, Irfan M, Siddique F, Arshad V, Zubairi ABS. Factors predicting in-hospital mortality among patients admitted with community acquired pneumonia at a tertiary care hospital Karachi, Pakistan. Clin Respir J. 2020 Apr;14(4):328-334. doi: 10.1111/crj.13137. Epub 2020 Jan 2. PMID 31863551
- [Result] Elsener C, Beeler PE, Battegay E, Bello B, Thienemann F. Risk Factors of In-Hospital Mortality in Patients Treated for Pneumonia at a Tertiary Care Centre in Switzerland. Respiration. 2020;99(8):637-645. doi: 10.1159/000508666. Epub 2020 Jul 7. PMID 32634800
- [Result] Li HY, Guo Q, Song WD, Zhou YP, Li M, Chen XK, Liu H, Peng HL, Yu HQ, Chen X, Liu N, Lu ZD, Liang LH, Zhao QZ, Jiang M. Modified IDSA/ATS Minor Criteria for Severe Community-Acquired Pneumonia Best Predicted Mortality. Medicine (Baltimore). 2015 Sep;94(36):e1474. doi: 10.1097/MD.0000000000001474. PMID 26356705
- [Result] Shoar S, Musher DM. Etiology of community-acquired pneumonia in adults: a systematic review. Pneumonia (Nathan). 2020 Oct 5;12:11. doi: 10.1186/s41479-020-00074-3. eCollection 2020. PMID 33024653
- [Result] 1. Somberg J. Harrisons, Princiole of Internal Medicine. 20th ed. LWW; 2005
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC7533148